CLINICAL TRIAL: NCT00199381
Title: An Open-Label Multicenter Study of the Continued Safety of Istradefylline (KW-6002) In Subjects With Parkinson's Disease Who Have Recently Completed One Year of Treatment With Istradefylline.
Brief Title: An Extension of Istradefylline in North American Parkinson's Disease Patients Who Have Completed Study 6002-INT-001
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Additional long-term safety data no longer needed
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6002-US-025
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Treatment with oral istradefylline (KW-6002) 20 or 40 mg once daily.
  Interventions: Drug: Istradefylline

INTERVENTIONS:
Drug: Istradefylline — Oral istradefylline (KW-6002) 20 or 40 mg once daily.
  Other Names: KW-6002

SUMMARY:
This is an, open-label, long-term safety extension for patients in North America who have completed the prior istradefylline study 6002-INT-001.

DETAILED DESCRIPTION:
Patients with Parkinson's disease with motor complications on levodopa therapy who completed the prior double-blind study 6002-INT-001 are eligible to enter into this long-term open safety study with a starting istradefylline dose of 20 or 40mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study 6002-INT-001
* Not of childbearing potential

Exclusion Criteria:

* Cancer within 5 years of enrollment
* ALT/AST levels > 2.5 times ULN

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Kyowa Pharmaceutical Inc., Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 study centers in the US and Canada recruited subjects from the initiation date (28 October 2005). Patients who had previously participated in Study 6002-INT-001 were eligible to participate in this follow-on safety study,and hence had been taking istradefylline for at least a year.
Pre-assignment Details: Subjects completing 6002-INT-001 immediately before entering the study had an interruption of study drug of 30 days or less. Qualifying subjects with an interruption of more than 30 days had their baseline visit after laboratory tests results were reviewed by the Investigator.
Period: Overall Study
Arm/Group | Single Arm
Started | 504
Completed | 0 (Premature study termination by the Sponsor.)
Not Completed | 504
Not completed — Withdrawal by Subject | 38
Not completed — Adverse Event | 73
Not completed — Protocol Violation | 6
Not completed — Lack of Efficacy | 27
Not completed — Not including due to early termination | 37
Not completed — Study termination by Sponsor | 323

BASELINE CHARACTERISTICS:
Population: 503 subjects took at least 1 dose of study drug
Arm/Group | Single Arm
Number analyzed (Participants) | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 244
  >=65 years | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 348
Region of Enrollment [Number; unit: participants] — 61 centers in the US and 12 centers in Canada recruited at least 1 subject
  participants
    United States | 401
    Canada | 102

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Adverse Events
Description: Investigation of the long-term tolerability and safety of istradefylline
Time Frame: Every 2 months up to 32 months
Population: Safety analysis set - all subjects who took at least one dose of study drug. 1 subject of the 504 enrolled did not take study drug and is not included in the safety analysis set.
Measure: Number; unit: participants
Arm/Group | Single Arm
Number analyzed (Participants) | 503
participants | 477

ADVERSE EVENTS:
Time Frame: Dosing to end of treatment.
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 201/503
Other Adverse Events (participants affected / at risk) | 276/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=503)
Parkinson's disease (Nervous system disorders) | 51 (55) — Worsening of Parkinson's disease
Syncope (Nervous system disorders) | 8 (8)
Cerebrovascular accident (Nervous system disorders) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Convulsion (Nervous system disorders) | 3 (3)
Lightheadedness (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Spinal cord compression (Nervous system disorders) | 2 (3)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (2)
Myasthenia gravis (Nervous system disorders) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (4)
Spondylosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extemity (Musculoskeletal and connective tissue disorders) | 1 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 9 (9)
Hip fracture (Injury, poisoning and procedural complications) | 8 (8)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Caustic injury (Injury, poisoning and procedural complications) | 1 (1)
Closed head injury (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Cellulitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (5)
Postoperative infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2)
Abscess jaw (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Diverticultis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Confusional state (Psychiatric disorders) | 10 (11)
Psychotic disorder (Psychiatric disorders) | 5 (5)
Delirium (Psychiatric disorders) | 4 (4)
Hallucination (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Markedly reduced dietary intake (Psychiatric disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (6)
Coronary artery disease (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (4)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress snydrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthenia (General disorders) | 3 (3)
Chest pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Drug interaction (General disorders) | 1 (1)
Gait abnormal (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4)
Colpocele (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1)
Urogenital prolapse (Reproductive system and breast disorders) | 1 (2)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Malignant hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (4)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Cardiac pacemaker revision (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Gangrenous cholecystitis (Hepatobiliary disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=503)
Nasopharyngitis (Infections and infestations) | 29
Upper respiratory tract infection (Infections and infestations) | 36
Urinary tract infection (Infections and infestations) | 47
Accident (Injury, poisoning and procedural complications) | 102
Arthralgia (Musculoskeletal and connective tissue disorders) | 63
Back pain (Musculoskeletal and connective tissue disorders) | 46
Parkinson's disease (Nervous system disorders) | 151 — Worsening of Parkinson's disease
Constipation (Gastrointestinal disorders) | 49
Nausea (General disorders) | 27
Asthenia (General disorders) | 29
Oedema peripheral (Cardiac disorders) | 41
Weight decreased (Investigations) | 35
Balance disorder (Nervous system disorders) | 38
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36
Dyskinesia (Nervous system disorders) | 136
Freezing phenomenon (Nervous system disorders) | 32
Lightheadedness (Nervous system disorders) | 33
Anxiety (Psychiatric disorders) | 40
Confusional state (Psychiatric disorders) | 29
Depression (Psychiatric disorders) | 54
Hallucination (Psychiatric disorders) | 69
Insomnia (Psychiatric disorders) | 49
Fatigue (General disorders) | 25
Headache (Nervous system disorders) | 26
Tremor (Nervous system disorders) | 35

LIMITATIONS AND CAVEATS:
The Sponsor decided to terminate the study early (not for safety reasons); as a result 323 subjects discontinued early. Mean duration of therapy was 18.7 months (0.4 to 31.4 months); median duration was 21.0 months. Total exposure 767 subject years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No